CLINICAL TRIAL: NCT07050966
Title: Comparative Effects of Maitland's Rotation Mobilization and Mulligan's Spinal Mobilization With Leg Movement on Lumbar Radiculopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/77
Record Dates: First submitted 2025-05-28; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Lumbar Radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Group A:
  * Mulligan Mobilization Technique: Spinal Mobilization with Leg Movement (3 reps, 3 sets)
  * Neurodynamic Mobilization (1 set, 3 reps)
  Interventions: Procedure: Group A (Active Comparator) 1. Mulligan's Spinal Mobilization with Leg Movement (SMWLM) 2.Lower Limb Neurodynamic Mobilization
- Group B (Experimental): Group B:
  Maitland Mobilization Technique; Lumbar rotation mobilization (3sets,3reps) Neurodynamic mobilization(1set,3reps)
  Interventions: Procedure: Group B (Experimental) 1. Maitland's Lumbar Rotation Mobilization 2.Lower Limb Neurodynamic Mobilization

INTERVENTIONS:
Procedure: Group A (Active Comparator) 1. Mulligan's Spinal Mobilization with Leg Movement (SMWLM) 2.Lower Limb Neurodynamic Mobilization — This group will receive Mulligan's Spinal Mobilization at the Lumbar Spine Region (L4-L5 level) along with Lower extremity movement (3 repetitions, 3 sets) followed by Neurodynamic Mobilization which will include slump technique (3 repetitions, 1 set). This protocol is given to the patient for a total of 6 sessions (1 session per day).
  Arms: Group A
Procedure: Group B (Experimental) 1. Maitland's Lumbar Rotation Mobilization 2.Lower Limb Neurodynamic Mobilization — This group will receive Maitland's Lumbar Rotation Mobilization at the Lumbar Spine Region (L4-L5 level) along with Lower extremity movement (3 repetitions, 3 sets) followed by Neurodynamic Mobilization which will include slump technique (3 repetitions, 1 set).This protocol is given to the patient for a total of 6 sessions (1 session per day).
  Arms: Group B

SUMMARY:
This study is a randomized control trial and the purpose of this study is to investigate and compare the effects of Maitland's rotation mobilization and Mulligan's spinal mobilization with leg movement (SMWLM) on lumbar radiculopathy patients.

DETAILED DESCRIPTION:
This study aims to combine the two separately established treatments techniques of mobilizations on patients with lumbar radiculopathy to find out which of the two has long lasting effects on:

1. Pain
2. Range of motion
3. Functional mobility

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years

  * Both Males and Females
  * Participants with a diagnosis of chronic (≥3 months) lumbar unilateral radiculopathy referred from Fauji Foundation Hospital, Rawalpindi
  * NPRS score of > 5 and < 8

Exclusion Criteria:

* Diagnosis of other back conditions (e.g. failed back surgery syndrome, spondylosis, spondylolisthesis, and spinal stenosis, non-specific low back pain, and fracture)

  * Non ambulant/wheelchair-bound or having cauda equina syndrome
  * Patient taking anticoagulants
  * Pregnant Females

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Lumbar Radiculopathy Pain | This protocol is given to the patient for a total of 6 sessions. NPRS is taken at the 1st, 3rd and 6th sessions respectively during the course of the treatment protocol.
  It will be measured using Numeric Pain Rating Scale (NPRS). Subjects select a number ranging from 0-10 according to their intensity of pain where '0' indicates no pain while '10' indicates worst pain experienced.
Range of Motion | This protocol is given to the patient for a total of 6 sessions. SLR Range is taken at the 1st, 3rd and 6th sessions respectively during the course of the treatment protocol.
  Universal goniometer is used to measure Straight Leg Raise Range (SLR) of the patient. Patient is positioned in supine with the knee straight. Axis of goniometer is aligned with the greater trochanter of the femur; stationary arm is kept parallel to the femur and moving arm is aligned with long axis of femur. Patient is then asked to flex the hip joint, keeping the knee straight, to the maximum range without pain, subsequently aligning moving arm of the goniometer. Angle of flexion is then recorded from the goniometer and documented.
Functional Status | This protocol is given to the patient for a total of 6 sessions. ODI Score is taken at the 1st, 3rd and 6th sessions respectively during the course of the treatment protocol.
  It is measured using Oswestry Disability Index Questionnaire (ODI-Q). The ODI-Q is a questionnaire used to assess an individual's ability to perform daily activities and functional tasks. It comprises of total 10 questions and patients rate their ability to perform each activity on a scale from 0 (unable to perform) to 5 (able to perform without difficulty). Each question has a maximum score of 5. The total maximum score is 50 which can change according to the number of total questions applicable to the respective patient. The obtained score is divided by the total score and multiplied by 100, giving a percentage as a result. Higher scores indicate better functional ability.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan